CLINICAL TRIAL: NCT02458469
Title: Pathogenesis of Sleep Disordered Breathing in Spinal Cord Injury Patients
Brief Title: Role of Enhancing Serotonin Receptors Activity for Sleep Apnea Treatment in Patients With SCI
Acronym: REST-SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NURC-062-12S; 1IK2CX000547 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injury; Sleep Disordered Breathing
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea Syndromes | interventions — Buspirone; Trazodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Buspirone (Active Comparator): This drug will be taken for two week period
  Interventions: Drug: Buspirone
- Trazodone (Active Comparator): This drug will be taken for two week period
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): A placebo pill will be taken at bed time for two week period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — The initial dose of Buspirone is 15 mg daily (7.5 mg bid.). To achieve an optimal therapeutic response, at intervals of 2 to 3 days the dosage may be increased 5 mg per day until a maximum dose 30mg/day is reached.
  Arms: Buspirone
Drug: Trazodone — 100 mg dose before bed-time
  Arms: Trazodone
Drug: Placebo — One placebo pill before bed-time
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at the effect of exciting using drugs to target a specific pathway in the body, that relies on a natural chemical the body produces called 'serotonin', in patients with spinal cord injury (SCI) during sleep. During this part of the study participants will be asked to take buspirone (Buspar) (15-50mg per day), trazodone (100mg per day) and a placebo in a random fashion, each for a 2 week period (drug period) of time followed by two weeks without drugs (washout period). The drugs will not be taken all at the same time, but each will be taken separately for two weeks followed by a night study to look at the effect the medication/placebo pill has on the way the body responds during sleep.

DETAILED DESCRIPTION:
Randomized placebo controlled cross-over study. Each subject will be studied on three separate occasions: (1) Buspirone vs. Trazodone vs. placebo for 2 weeks; the patients will be blinded to whether they are taking trazodone or placebo; buspirone cannot be blinded because it is dosed twice a day and is up titrated during the two weeks of administration. The initial dose of Buspirone is 15 mg daily (7.5 mg bid.). To achieve an optimal therapeutic response, at intervals of 2 to 3 days the dosage may be increased 5 mg per day until a maximum dose 30mg/day is reached. After the two week treatment a sleep study will be repeated. Trazodone will be given at 100 mg dose before bed-time. (2) Cross over medication for two weeks will be followed by a second sleep study followed by two weeks washout. (3) Cross over medication for two weeks will be followed by another sleep study. To assess the clinical effect of the drug on breathing during sleep a qualitative polysomnography will be performed for 2 hours the same night after taking the drug/placebo. This will allow the determination of ventilatory changes and the determination of the number of respiratory events (apnea/hypopnea index).

ELIGIBILITY:
Inclusion Criteria:

* Adults with SCI (>6months after spinal cord injury) at the T6 level/above

Exclusion Criteria:

* Pregnant and lactating females
* Heart failure, vascular disease, or stroke
* Advanced chronic obstructive pulmonary disease (COPD), liver disease, and chronic kidney disease
* BMI >38 kg/m2
* Mechanical ventilation dependence
* The following medications are not allowed (potential interaction with buspirone or inhibition of the CYP3A4 system):

  * cimetidine
  * ketoconazole
  * ritonavir
  * itraconazole
  * erythromycin
  * diltiazem
  * verapamil
  * Monoamine oxidase (MAO) inhibitors [such as Marplan, Nardil, Parmate, Emsam]
  * Other prohibited concomitant medications include haloperidol, trazodone, or triazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulghani Sankari, MD PhD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the primary site at John D. Dingell VA Medical Center.
Pre-assignment Details: Of 150 available, 15 participants were enrolled. Of the 15 enrolled, 11 started the study protocol.
Groups:
- Placebo->Buspirone->Trazodone: Participants first received a placebo taken once daily for two weeks. After a washout period of two weeks, the participants then received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks. After another washout period of two weeks, participants received trazodone (100 mg) once daily for two weeks.
- Placebo->Trazodone->Buspirone: Participants first received a placebo taken once daily for two weeks. After a washout period of two weeks, the participants then received trazodone (100 mg) once daily for two weeks. After another washout period of two weeks, participants received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks.
- Buspirone->Trazodone->Placebo: Participants first received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks. After a washout period of two weeks, the participants then received trazodone (100 mg) once daily for two weeks. After another washout period of two weeks, participants received a placebo taken once daily for two weeks.
- Buspirone->Placebo->Trazodone: Participants first received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks. After a washout period of two weeks, the participants then received a placebo taken once daily for two weeks. After another washout period of two weeks, participants received trazodone (100 mg) once daily for two weeks.
- Trazodone->Placebo->Buspirone: Participants first received trazodone (100 mg) once daily for two weeks. After a washout period of two weeks, the participants then received a placebo taken once daily for two weeks. After another washout period of two weeks, participants received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks.
- Trazodone->Buspirone->Placebo: Participants first received trazodone (100 mg) once daily for two weeks. After a washout period of two weeks, the participants then received buspirone taken twice daily (7.5 - 15 mg) on an increasing scale for two weeks. After another washout period of two weeks, participants received a placebo taken once daily for two weeks.
Period: First Intervention (2 Weeks)
Arm/Group | Placebo->Buspirone->Trazodone | Placebo->Trazodone->Buspirone | Buspirone->Trazodone->Placebo | Buspirone->Placebo->Trazodone | Trazodone->Placebo->Buspirone | Trazodone->Buspirone->Placebo
Started | 3 | 2 | 3 | 0 | 1 | 2
Completed | 2 | 2 | 2 | 0 | 1 | 2
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Period: First Washout (2 Weeks)
Arm/Group | Placebo->Buspirone->Trazodone | Placebo->Trazodone->Buspirone | Buspirone->Trazodone->Placebo | Buspirone->Placebo->Trazodone | Trazodone->Placebo->Buspirone | Trazodone->Buspirone->Placebo
Started | 2 | 2 | 2 | 0 | 1 | 2
Completed | 2 | 2 | 2 | 0 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Placebo->Buspirone->Trazodone | Placebo->Trazodone->Buspirone | Buspirone->Trazodone->Placebo | Buspirone->Placebo->Trazodone | Trazodone->Placebo->Buspirone | Trazodone->Buspirone->Placebo
Started | 2 | 2 | 2 | 0 | 1 | 2
Completed | 2 | 2 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Washout (2 Weeks)
Arm/Group | Placebo->Buspirone->Trazodone | Placebo->Trazodone->Buspirone | Buspirone->Trazodone->Placebo | Buspirone->Placebo->Trazodone | Trazodone->Placebo->Buspirone | Trazodone->Buspirone->Placebo
Started | 2 | 2 | 2 | 0 | 1 | 1
Completed | 2 | 2 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | Placebo->Buspirone->Trazodone | Placebo->Trazodone->Buspirone | Buspirone->Trazodone->Placebo | Buspirone->Placebo->Trazodone | Trazodone->Placebo->Buspirone | Trazodone->Buspirone->Placebo
Started | 2 | 2 | 2 | 0 | 1 | 1
Completed | 2 | 2 | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Buspirone (7.5-15 mg) or Trazodone (100 mg) or Placebo tablet
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: CO2 Reserve (Delta-PETCO2-AT)
Description: Randomized placebo-controlled cross-over study. Each subject was studied on three separate occasions: (1) Buspirone vs. Trazodone vs. placebo for 2 weeks; After the two-week treatment a noninvasive nasal mechanical ventilation study was repeated to determine the hypocapnic apneic threshold. (2) Cross over medication for two weeks was followed by a second noninvasive nasal mechanical ventilation study to determine the CO2 reserve (Delta-PETCO2-AT) and hypocapnic apneic threshold followed by two weeks washout. (3) Cross over medication for two weeks was followed by another sleep study to determine the hypocapnic apneic threshold.
Time Frame: Two weeks
Population: Only 8 of the 15 enrolled participants finished all three medication arms (placebo, buspirone, trazodone) and were used in the final analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buspirone | Trazodone | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mmHg | -3.6 (0.9) | -2.5 (1.0) | -1.8 (1.5)
Statistical Analysis 1: Comparison: Buspirone vs Trazodone vs Placebo; Test type: Superiority; p = 0.019, ANOVA
Statistical Analysis 2: Comparison: Buspirone vs Placebo; Test type: Superiority; p = 0.015, Student-Newman-Keuls Method
Statistical Analysis 3: Comparison: Trazodone vs Placebo; Test type: Superiority; p = 0.231, Student-Newman-Keuls Method

2. Secondary Outcome: Apnea-Hypopnea Index (AHI)
Description: Randomized placebo-controlled cross-over study. Each subject was studied on three separate occasions: (1) Buspirone vs. Trazodone vs. placebo for 2 weeks; After the two-week treatment a polysomnogram (PSG) study was repeated to determine the AHI. (2) Cross over medication for two weeks was followed by a second PSG to determine the AHI followed by two weeks washout. (3) Cross over medication for two weeks was followed by another sleep study to determine the AHI.
Time Frame: Two weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events/Hour
Arm/Group | Buspirone | Trazodone | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Events/Hour | 48.7 (21.4) | 40.0 (23.9) | 45.2 (23.2)
Statistical Analysis 1: Comparison: Buspirone vs Trazodone vs Placebo; Test type: Superiority; p = 0.749, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the two-week interventions during which the participants were taking Buspirone, Trazodone, or placebo.
Description: Of the 11 participants who started the study protocol, 10 received Buspirone, 9 received Trazodone, and 9 received a placebo due to participant withdrawal and physician removal.
Arm/Group | Buspirone | Trazodone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 3/10 | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=10) | Trazodone (N=9) | Placebo (N=9)
Suicidal Thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=10) | Trazodone (N=9) | Placebo (N=9)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
* The sample size is small and the majority are males, therefore findings from this study may not be applicable to the general population
* The study required heavy instrumentation which may have affected natural sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT02458469/Prot_SAP_000.pdf